CLINICAL TRIAL: NCT07360080
Title: Long-Term Outcomes of Participants Treated With Teplizumab in Routine Clinical Care
Brief Title: Long-Term Outcomes of Teplizumab in Routine Clinical Care
Acronym: AL1GN
Status: Not yet recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18569; U1111-1317-7939 (Other: ICTRP)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Stage 2 Type 1 Diabetes (T1D) who received Teplizumab
  Interventions: Drug: Teplizumab

INTERVENTIONS:
Drug: Teplizumab — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practice.

SUMMARY:
This is an observational, prospective cohort study designed to evaluate the outcomes after teplizumab treatment in participants with Stage 2 Type 1 Diabetes (T1D) for delaying the onset of Stage 3 T1D. The study will monitor participants receiving teplizumab as part of routine clinical care across multiple sites. Additionally, patient-reported outcomes (PROs) will be evaluated to further assess the treatment's impact on participant's quality of life including emotional and psychosocial aspects associated with T1D. This approach will provide a more comprehensive understanding of how the treatment performs over time and across diverse patient populations, providing valuable insights into the sustained effects of teplizumab and offering a real world picture of its impact on the long-term management of T1D.

DETAILED DESCRIPTION:
Enrolled participants will be followed for up to 10 years depending on the time the participants are included after initiating teplizumab treatment.

ELIGIBILITY:
Inclusion Criteria -

* Participants who have received at least 1 teplizumab infusion within 6 weeks prior to enrollment.
* Participants must have a confirmed diagnosis of Stage 2 T1D according to the treating physician at the time of the first infusion of teplizumab.

(Note: Participants who progress to Stage 3 T1D by Week 6 will still be eligible, provided they were in Stage 2 at the time of the first teplizumab infusion.)

• Participants (or their legal guardians, as applicable) who provide appropriate written or electronic informed consent/assent as applicable for the age of the participant and as per local regulations.

Exclusion Criteria -

* Participants who had participated in a previous clinical trial for teplizumab.
* Participants enrolled in a clinical trial within 6 months prior to study enrollment.

(Note: Participants enrolled in other observational studies may be included.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Stage 2 T1D who have received at least 1 teplizumab infusion within 6 weeks prior to enrollment. Approximately 1000 participants, in 85 sites across 19 countries will be enrolled over 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2035-10-29 (Estimated); Study Completion 2035-10-29 (Estimated)

PRIMARY OUTCOMES:
Time from teplizumab infusion start to the onset of Stage 3 T1D | From start of infusion to maximum of 10 years

SECONDARY OUTCOMES:
Proportion of participants who complete teplizumab treatment course | Up to end of infusion, maximum of 5 years
Number of participants with adverse events during the infusion period | Till 6 weeks post last infusion, maximum of 5 years
Number of participants with adverse events of special interest and serious adverse events | From 6 weeks post last infusion through the follow-up, maximum of 10 years
Number of participants with T1D-related complications | From infusion up to end of study, maximum of 10 years
  Including but not limited to the following: diabetic ketoacidosis, severe hypoglycemia, retinopathy, nephropathy, neuropathy, cardiovascular events
Glycemic control assessment values | From baseline through follow-up, maximum of 10 years
Change from baseline in glycated hemoglobin (HbA1c) | From baseline through follow-up, maximum of 10 years
Proportion of participants achieving target HbA1c ≤ 6.5% | From baseline through follow-up, maximum of 10 years
Proportion of participants using home glycemic control assessments (eg, SMBG, CGM) | From baseline through follow-up, maximum of 10 years
Proportion of participants using glycemic control assessments in-clinic (eg, OGTT, FPG, MMTT, RPG) | From baseline through follow-up, maximum of 10 years
Mean change from baseline in Time in range (TIR) (70 to 180 mg/dL [3.9 to 10 mmol/L]) | From baseline through follow-up, maximum of 10 years
  CGM reading 70 to 180 mg/dL [3.9 to 10 mmol/L]
Mean change from baseline in Time in tight range (TITR) (70 to 140 mg/dL [3.9 to 7.8 mmol/L]) | From baseline through follow-up, maximum of 10 years
  CGM reading 70 to 140 mg/dL [3.9 to 7.8 mmol/L]
Mean change from baseline in Time above tight range (TATR): >140 mg/dL (>7.8 mmol/L) | From baseline through follow-up, maximum of 10 years
  CGM reading >140 mg/dL (>7.8 mmol/L)
Mean change from baseline in Time above range (TAR): >180 mg/dL (>10 mmol/L) | From baseline through follow-up, maximum of 10 years
  CGM reading >180 mg/dL (>10 mmol/L)
Mean change from baseline in Time above range (TAR): >250 mg/dL (>13.9 mmol/L) | From baseline through follow-up, maximum of 10 years
  CGM reading >250 mg/dL (>13.9 mmol/L)
Mean change from baseline in Time below range (TBR): <70 mg/dL (<3.9 mmol/L) | From baseline through follow-up, maximum of 10 years
  CGM reading <70 mg/dL (<3.9 mmol/L)
Mean change from baseline in Time below range (TBR): <54 mg/dL (<3.0 mmol/L) | From baseline through follow-up, maximum of 10 years
  CGM reading <54 mg/dL (<3.0 mmol/L)
Mean change from baseline in within-day glucose coefficient of variation | From baseline through follow-up, maximum of 10 years
Mean change from baseline in between-day glucose coefficient of variation | From baseline through follow-up, maximum of 10 years
Proportion of participants using insulin during the study period | Up to end of study, maximum of 10 years
  Continuous subcutaneous insulin infusion, insulin pump, or pump integrated with an automated insulin delivery system
Proportion of participants using other glucose lowering therapies during the study period | Up to end of study, maximum of 10 years
Change in EuroQol 5-Dimensions (EQ-5D) scores in adult and pediatric participants | From the first posttreatment visit after the last teplizumab infusion through follow-up, for a maximum of 10 years
Change in Hospital Anxiety and Depression Scale (HADS) scores in adult participants | From the first posttreatment visit after the last teplizumab infusion through follow-up, for a maximum of 10 years
Change in World Health Organization-Five Well-Being Index (WHO-5) scores in pediatric participants | From the first posttreatment visit after the last teplizumab infusion through follow-up, for a maximum of 10 years
Change in Diabetes Distress Scale (DDS) scores in adult participants | From the time of Stage 3 T1D confirmation through follow-up, for a maximum of 10 years
Change in Hypoglycemia Fear Survey-II (HFS-II) scores in adult and pediatric participants | From the time of Stage 3 T1D confirmation through follow-up, for a maximum of 10 years
Annualized rate of hospitalizations due to T1D related disease and complications | Up to end of study, maximum of 10 years
Annualized rate of emergency room visits related to T1D related disease and complications | Up to end of study, maximum of 10 years

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.